CLINICAL TRIAL: NCT03564912
Title: Prospective Study on the Efficacy and Safety of 2 Week or 3 Week Xelox Regimen for Adjuvant Chemotherapy in Colorectal Patients After Surgery
Brief Title: Prospective Study on the Efficacy and Safety of 2 Week or 3 Week Xelox Regimen for Adjuvant Chemotherapy in CRC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, director, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangU020
Record Dates: First submitted 2018-05-27; First posted 2018-06-21 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2 week group (Experimental)
  Interventions: Drug: Capecitabine Oral Tablet [Xeloda]
- 3 week group (Active Comparator)
  Interventions: Drug: Capecitabine Oral Tablet [Xeloda]

INTERVENTIONS:
Drug: Capecitabine Oral Tablet [Xeloda] — 2 week group: capecitabine 1000mg/m2 d1-10; oxaliplatin 85mg/m2; q2w 3 week group: capecitabine 1000mg/m2 d1-14; oxaliplatin 130mg/m2; q3w
  Other Names: oxaliplatin

SUMMARY:
This study select the diagnosis of postoperative colorectal cancer patients with stage II/III to adjuvant chemotherapy, and received 2 weeks and 3 weeks xelox adjuvant treatment process until disease progression or patients died or lost to follow-up. To analyze the difference in efficacy and safety of xelox in 2 weeks and 3 weeks of postoperative adjuvant therapy for colorectal cancer, so as to find a better postoperative adjuvant treatment model.

ELIGIBILITY:
Inclusion Criteria:

* Carcinoma of the intestine confirmed histologically or cytologically
* Radical surgical resection was performed after diagnosis and the post operative stages were high-risk II or III patients
* The ECOG PS score less than or equal to 2 points
* No chemotherapy of any kind has been performed in the past
* Neutrophils acuity 1.5x10e9/L, platelets more than 100x10e9/L, college blood red protein more than 9g/dL
* liver function transaminase is less than or equal to 2.5 ULN, alkaline phosphatase is less than 2.5 ULN, and total bilirubin is less than 1.5 ULN

Exclusion Criteria:

* Patients with unresectable CRC
* Patients who have any form of chemotherapy before
* Participating in or having participated in clinical studies of other drug
* Patients have second primary malignant tumors of have other malignant tumors in the past five years
* There is evidence of allergic reaction to drugs in this study
* A history of ischemic heart disease in the past 1 year or patients with high risk factors for heart failure, or uncontrolled arrhythmias
* Severe active inflammation, including tuberculosis and HIV
* Long-term immunization or hormone therapy, except hormone replacement therapy at physiological dose
* Drug or alcohol addiction
* Get pregnant or breastfeed
* The investigator considers that the patient is not suitable for this clinical study due to any clinical or laboratory abnormalities or compliance problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
DFS | through study completion, an average of 1 year
  disease free survival

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 weeks
  toxicity difference of two groups

CONTACTS AND LOCATIONS:
Locations (1):
- First afflicated hospital of zhejiang university, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhang H, Wang D, Tong Z, Xiang T, Zhu X, Liu L, Zheng Y, Zhao P, Fang W, Chen W. Biweekly CAPOX versus triweekly CAPOX in the adjuvant therapy of post-surgery CRC: A randomized controlled trial. PLoS One. 2025 Jul 11;20(7):e0313472. doi: 10.1371/journal.pone.0313472. eCollection 2025. PMID 40644418